CLINICAL TRIAL: NCT04136847
Title: A Single-Center Trial to Evaluate the Efficacy and Tolerability of the SkinPen on Male and Female Subjects' Dorsal Hands as a Treatment for Signs of Hand Aging
Brief Title: Study to Evaluate the Efficacy and Tolerability of the SkinPen on Male and Female Subjects' Dorsal Hands as a Treatment for Signs of Hand Aging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 19 the Study did not start enrolling
Sponsor: Bellus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bellmed003
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Aging
Keywords: Signs of Hand Aging

STUDY DESIGN:
Intervention Model Description: At least twenty three (23) qualified and consenting subjects treated with 4 Skinpen microneedling treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hand Aging (Experimental): Microneedling treatment of the dorsum of the hands
  Interventions: Device: SkinPen Precision

INTERVENTIONS:
Device: SkinPen Precision — Surgical instrument motors and accessories/attachments/Hydrogel

SUMMARY:
Microneedling is a relatively new, minimally invasive technique originally developed for skin rejuvenation. Controlled micro-injury to the dermis via the application of several small needles connected to a motorized device stimulates the wound healing process, resulting in the formation of new tissue and blood vessels. The SkinPen by Bellus Medical is an FDA-cleared microneedling device proven to improve the appearance of acne scars This study evaluates the clinical performance of the SkinPen device for the treatment of signs of aging on the back of the hand.

DETAILED DESCRIPTION:
SkinPen microneedling treatment of dorsal hand skin This is a single-site, non-randomized, non-controlled study designed to follow at least twenty

three (23) qualified and consenting subjects treated with 4 Skinpen microneedling treatments. The sample size determination of this study is based on the recommendations of the sponsor. These patients will be treated four times over the dorsum of the hand from the wrist to the knuckles each month for four months, followed by two follow-up visits at 1-month and 3-months post-treatment. The acute effects of microneedling will be determined by subjective and objective analysis using standard and close-up photography. Additionally, the effects of this treatment will be analyzed at 1-month and 3-month post-treatment through clinician and subject assessments.

Subjects will be identified from Dr. Jeffrey Kenkel's clinical practice at the University of Texas Southwestern Medical Center. Subjects will be numbered sequentially in the order in which they qualify for entry into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 50 to 75 years of age having general good health.
2. Individuals deemed by the Investigator, visually, to have signs of hand aging (presence of skin laxity, age spots, trophic changes) on the dorsum of the hand.. Also, Subjects would have to be willing to undergo correction of these signs of aging.
3. Individuals willing to withhold aesthetic therapies to the areas of the hand being treated or judged to potentially impact results by the Investigator (e.g. soft tissue fillers and/or any resurfacing procedures, botulinum toxin, injectable fillers, microdermabrasion, IPL (intense pulsed light), peels, laser treatments, and tightening treatments, etc.) for the duration of the study. Waxing and threading is allowed but not laser hair removal.
4. Individuals that are willing to provide written informed consent
5. Individuals willing to sign a photography release.
6. Willingness to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.
7. Women of child bearing potential agree to take a urine pregnancy test at the Baseline visit and 3-months post-treatment or when deemed by Investigator and/or Sponsor. This may be changed to a monthly pregnancy test at the Sponsor's discretion. Women who are of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the baseline visit. Women must be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   * Postmenopausal for at least 12 months prior to study;
   * Without a uterus and/or both ovaries;
   * Bilateral tubal ligation at least 6 months prior to study enrollment.

Exclusion Criteria:

1. Individuals diagnosed with known allergies to general skin care products.
2. Individuals who have presence of an active systemic or local skin disease that may affect wound healing.
3. Individuals who have severe solar elastosis.
4. Individuals with sensitivity to topical lidocaine.
5. Individuals who have physical or psychological conditions unacceptable to the Investigator.
6. Individuals who have a recent history of significant trauma to the areas to be treated (< 6 months).
7. Individuals who have significant scarring in the area(s) to be treated.
8. Individuals who have a recent or current history of inflammatory skin disease, infection or unhealed wound.
9. Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g. Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyositis, etc.).
10. Individuals who currently have or have a history of hypertrophic scars, or keloid scars.
11. Individuals who currently have cancerous or pre-cancerous lesions in the areas to be treated and/or with a history of skin cancer.
12. Individuals who have the inability to understand instructions or to give informed consent.
13. Individuals who have had microdermabrasion or glycolic acid treatment to the treatment area(s) within one month prior to study participation or who will have this treatment during the study.
14. Individuals who have a history of chronic drug or alcohol abuse.
15. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
16. Individuals who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
17. Individuals who are current smokers or have smoked in the last five years.
18. Individuals who have a history of the following cosmetic treatments in the area(s) to be treated:

    * Skin tightening procedure within the past year;
    * Injectable filler of any type within the past:

      * 12 months for Hyaluronic acid fillers (e.g. Restylane)
      * 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)
      * 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra)
      * Ever for permanent fillers (e.g. Silicone, ArteFill)
    * Neurotoxins within the past three months;
    * Ablative resurfacing laser treatment;
    * Non-ablative, rejuvenative laser or light treatment within the past six months;
    * Surgical dermabrasion;
    * Had a chemical peel or dermabrasion, of the dorsum of the hand within four weeks
19. Individuals with a history of using the following prescription medications:

    * Accutane or other systemic retinoids within the past six months;
    * Topical Retinoids within the past two weeks;
    * Prescription strength skin lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA and polyhydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within four months;
    * Any anti-wrinkle, skin lightening devices, or any other device or topical or systemic medication known to affect skin aging or dyshcromia (devices containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, gigawhite, lemon juice extract (topically), emblica extract, etc.) within two weeks;
    * Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use); and/or
    * Psychiatric drugs that in the Investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
20. Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
21. Individuals having a health condition and/or pre-existing or dormant dermatologic disease on the body (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
22. Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
23. Individuals with an uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
24. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
25. Individuals who have observable suntan, nevi, excessive hair, etc. or other dermal conditions on the back of the hand that might influence the test results in the opinion of the Investigator or designee.
26. Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other cosmetic treatments to the treatment area; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments).
27. Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than three months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Aesthetic Assessment of change | 6 months
  Clinician's global aesthetic improvement assessment (CGAIS) , a 5 point grading scale where 1 is ''Very Much Improved'' and 5 is ''Worse''
Aesthetic Assessment | 6 months
  Subject's global aesthetic improvement assessment (CGAIS) , a 5 point grading scale where 1 is ''Very Much Improved'' and 5 is ''Worse''

SECONDARY OUTCOMES:
Adverse Events | 6 months
  Monitoring of adverse events throughout the course of the study.
Skin density | 6 months
  Ultrasound Imaging System
Skin Firmness | 6 months
  BTC 2000
Assessments of aging signs | 6 months
  Measurements acquired by the VISIA Complexion Analysis System
Treatment satisfaction assessment | 6 months
  Patient Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UTSW
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States